CLINICAL TRIAL: NCT05642429
Title: A Phase I, Randomized, Double-Blind Study to Evaluate Safety and Tolerability of Amyloid-β Vaccine, AV-1959D, in Patients With Early Alzheimer's Disease.
Brief Title: Study of AV-1959D, an Amyloid Beta Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Molecular Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Clinartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IMM-AV1959D-101; R01AG074983 (NIH)
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AV-1959D 500 μg (Active Comparator)
  Interventions: Biological: AV-1959D
- AV-1959D 1000 μg (Active Comparator)
  Interventions: Biological: AV-1959D
- AV-1959D 2000 μg (Active Comparator)
  Interventions: Biological: AV-1959D
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AV-1959D — Three doses of AV-1959D administered as a sterile suspension via intradermal injection
  Arms: AV-1959D 1000 μg; AV-1959D 2000 μg; AV-1959D 500 μg
Biological: Placebo — Three doses of Placebo administered as a sterile suspension via intradermal injection
  Arms: Placebo

SUMMARY:
Phase 1 clinical trial of AV-1959 amyloid-β vaccine for Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The Phase I study is a randomized, multicenter, double-blind, placebo-controlled study consisting of 3 sequential cohorts to determine the safety and tolerability of AV-1959D at three doses compared to a placebo in patients with early AD

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects from 60 to 85 years of age, both inclusive.
2. Mild cognitive impairment (MCI) due to Alzheimer's disease (AD), according to Albert et al., or mild AD dementia, according to McKhann et al., and must have the following:

   * Mini-Mental State Examination (MMSE) score from 22 to 30;
   * Clinical Dementia Rating (CDR) global score of 0.5 or 1.0.
3. A positive visual Aβ positron emission tomography (PET) scan. Previously obtained PET scan (within 24 months of screening) is permissible and must be submitted to the central imaging reader to confirm that study inclusion criteria are met.
4. Subjects on approved AD medications (e.g., acetylcholine esterase inhibitors, memantine) are required to be on a stable dose for a minimum 3 months before baseline and with no dosage adjustments expected during the study. Continuation of subjects with dose adjustments for approved AD medications during the study may be allowed after discussion between the Investigator and the Medical Monitor.
5. The subject has a reliable study partner who will accompany the patient to all clinic visits during the study and, in the Investigator's opinion, has frequent and sufficient contact with the subject as to be able to provide accurate information about the subject's cognitive and functional abilities.
6. The subject's sight and hearing (hearing aid permissible) are sufficient for compliance with the study procedures.
7. Signed informed consent form by the subject and study partner prior to study participation.

Exclusion criteria:

1. Participation in another investigational drug or device study or treated with an investigational drug within 30 days or 5 half-lives, whichever is longer, before dosing.
2. Prior administration of any amyloid-beta or tau immunotherapy (vaccine, antibody)
3. Magnetic resonance imaging (MRI) showing evidence of any of the following:

   * More than 1 lacunar infarct greater than 1.5 cm
   * Any territorial infarct, including acute or chronic, greater than 1.5 cm
   * Subjects who have a combined number of microbleeds and areas of leptomeningeal hemosiderosis (i.e., cumulative ARIA-H) on the MRI of > 5 (and should not include any disseminated leptomeningeal hemosiderosis)
   * Subjects who have a presence of any other significant cerebral abnormalities, including ARIA-E, as assessed in the screening MRI scan.
4. Contraindications for MRI scanning, including implanted metallic devices (e.g., non-MRI-safe cardiac pacemaker or neurostimulator; some artificial joints metal pins; surgical clips; or other implanted metal parts), or claustrophobia or discomfort in confined spaces.
5. Use of immunomodulatory or growth-stimulating factors such as systemic corticosteroids, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, GM-CSF, C-CSF, interferon (IFN), or interleukin-2 (IL-2) within 30 days prior to study entry.
6. Concurrent use of warfarin or other coumarin derivatives or a combination of acetylsalicylic acid and an anti-platelet agent (e.g., clopidogrel). Low dose of acetylsalicylic acid (≤81 mg per day) is allowed.
7. Parenteral use of immunoglobulin preparations, blood products, plasma derivatives.
8. Any serious illness requiring systemic treatment and/or hospitalization within 4 weeks prior to study entry.
9. Any major or unstable illness, including unstable ischemic cardiovascular disease, or require use of excluded medications.
10. History/evidence of clinically relevant pathology related to cardiovascular system, respiratory tract, gastrointestinal tract, endocrinology, immunology, hematology, or any other systemic disorder/major surgeries that in the opinion of the Investigator would confound the subject's participation and follow-up in the clinical study.
11. Subjects with insulin-dependent diabetes.
12. Cardiac arrhythmias or palpitations [e.g., supraventricular tachycardia, atrial fibrillation, frequent ectopy, or sinus bradycardia]. Cardiac conduction abnormalities to be specified including prolonged QT interval and bundle branch blocks.
13. Subjects with pre-existing autoimmune diseases.
14. A medical condition that in the opinion of the Investigator might be a contributing cause of cognitive impairment.
15. History/evidence of severe local or systemic reactions to vaccination or significant allergic reactions.
16. History of seizure disorder.
17. Any other medical, psychological, social condition or diagnostic test which, in the opinion of the Investigator and Medical Monitor may lead to screen failure or prevent the subject from fully participating in the study, represent a concern for study compliance, or constitute a safety concern to the subject.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs) | Baseline up to Week 28 weeks

SECONDARY OUTCOMES:
Number of participants with clinically significant changes in vital signs | Baseline up to Week 28
Number of participants with clinically significant changes in ECG results | Baseline up to Week 28
Number of participants with clinically significant changes in laboratory test | Baseline up to Week 28
Number of participants with clinically significant changes in physical examinations | Screening up to Week 28
Number of participants with clinically significant changes in neurological examinations | Screening up to Week 28
Number of participants with Vasogenic edema (ARIA-E) | Screening, Weeks 8 and 28
Number of participants with New cerebral ischemic or hemorrhagic events (ARIA-H) or associated symptoms | Screening, Weeks 8 and 28
Number of participants with Change from baseline in C-SSRS Score | Baseline, Weeks 12 and 28
Immunological outcome | Baseline and up to Week 28 post start of immunization with AV-1959D
  * Detection of possibly harmful autoreactive Th cell responses specific to Aβ.
  * Serum anti-Aβ antibodies concentrations.
  * Detection of Th cell responses specific to the MultiTEP platform.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Agadjanyan, PhD, Study Director — IMM
Locations (6):
- United States (6):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Hoag Memorial Hospital, Newport Beach, California
  - University of South Florida, Tampa, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Accel Research, Decatur, Georgia
  - Global Medical Institutes Princeton Medical Institute, Princeton, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided